CLINICAL TRIAL: NCT00498238
Title: The Effect of Levothyroxine on Arterial Stiffness and Lipid Profile in Patients
Brief Title: The Effect of Levothyroxine on Arterial Stiffness and Lipid Profile in Patients With Subclinical Hypothyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ronit1
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2007-07-09 (Estimated); Status verified 2007-07

CONDITIONS: Subclinical Hypothyroidism
Keywords: Arterial stiffness, Augmentation index, Subclinical Hypothyroidism
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levothyroxine

SUMMARY:
We evaluated the effect of levothyroxine in subclinical hypothyroidism (SCH) on arterial stiffness, lipid profile and inflammation. Thirty-four patients with SCH were included. Patients were treated with levothyroxine for 7 months. Arterial stiffness was evaluated by Augmentation index (AIx). After accomplishing euthyroidism, the AIx decreased from 8.3±17.2 to 6.5±14.3(P<0.01) and AIx percentage decreased from36.2 11.5 ± to 9.1±33.2 (P =0.03). Systolic blood pressure decreased from 20±134.7 to mmHg 13.7±127.6 (P<0.01). No significant improvement was found in other parameters. In patients whose AIx's decreased, LDL-cholesterol levels decreased by 37.1±-15.5 mg/dl compared to the patients whose AIx's didn't decrease and LDL-cholesterol increased by 57.4±24.1 mg/dl (P=0.057). We concluded that in patients suffering from SCH, treatment with levothyroxine had a significant beneficial effect on arterial stiffness and systolic blood pressure and no effect on lipid profile or inflammation.

DETAILED DESCRIPTION:
Subclinical hypothyroidism (SCH) is a disorder characterized by high levels of thyrotropin (thyroid stimulating hormone (TSH)), accompanied by normal levels of thyroxine (T4). There is most probably an association between SCH and cardiovascular disease, however the relationship between SCH and cardiovascular morbidity and mortality is still in debate.

Hak et al. and Walsh et al. found that patients with SCH have increased risk for ischemic heart disease. Female smokers over 50 years, with TSH levels above 10 mU/L, were at a higher risk. However, a study conducted by Rodondi et al. did not find that SCH increases the risk for cardiac ischemia, peripheral vascular disease or cerebrovascular disease.

Among the risk factors for atherosclerosis in patients with SCH are hypertention, atherogenic lipid profile, high levels of c-reactive protein (CRP), changes in the clotting system, endothelial dysfunction and increased arterial stiffness.

Studies have shown that patients with SCH suffer from increased arterial stiffness and endothelial dysfunction. One of the non invasive techniques to evaluate arterial stiffness is pulse wave analysis (PWA). PWA gives information of blood pressure at the aortic site rather than more peripherally. Recently, calculated AIx was suggested as an independent risk marker for cardiovascular adverse events. Obuobie et al. analyzed the pressure wave velocity in 12 patients with overt hypothyroidism treated with levothyroxine. They concluded that hypothyroid patients treated with levothyroxine had a decrease in their arterial stiffness after treatment, although no difference in the lipid profile was found.

Taddei et al. showed that patients with SCH are characterized by endothelial dysfunction resulting from a reduction in nitric oxide (NO); this alteration was partially independent of dyslipidemia and reversed by levothyroxine treatment.

The aim of this study was to assess the effect of levothyroxine treatment on blood pressure, lipid profile, highly sensitive CRP (hs- CRP) and arterial stiffness in patients with SCH. Whether SCH is a "laboratory" disease only or it affects blood vessels is a question still in controversy. We do not know yet if levothyroxine therapy will reverse some of the "silent" problems of SCH.

Methods

Patients Thirty four patients with laboratory evidence of subclinical hypothyroidism (TSH levels 4-25 mU/L and normal T4 values) in at least two following tests (one month apart from each other) were recruited from an endocrinology outpatient clinic for this study.

The protocol was approved by the local Helsinki Committee for experiments on Humans and all patients gave informed consent. The exclusion criteria were recent (less than 6 months) myocardial infarction, cerebrovascular event or angiography with stent placement, serious infection in the month before recruitment, any use of contrast media in the last 6 months, loss of more than 5% of body weight during the last 6 months, cardiac arrhythmias, ejection fraction of less than 40%, active malignant diseases, previous thyroid disease and pregnancy.

Study design The patients were treated with levothyroxine (Eltroxin, Glaxo) at a starting dose of 50 mcg per day. The follow up was conducted in the Research and Development unit, Assaf Harofeh Medical Center at 1, 4 and 7 months post dosing. In patients who did not achieve normalization of TSH, the dose of levothyroxine was increased to 100 mcg per day.

At each visit the patients underwent a physical examination including blood pressure, pulse and weight. Blood pressure was measured while the patient was in a recumbent position. Blood was drawn for TSH, Hemoglobin, renal and liver function, total cholesterol, high density lipoprotein-cholesterol (HDL- cholesterol), triglycerides (TG), oxidized low density lipoprotein (ox-LDL) and hs- CRP. LDL-cholesterol was calculated and arterial stiffness was assessed. The patients' medication regimen was not changed throughout the study period.

Arterial stiffness Assessment of arterial stiffness was performed by a noninvasive technique using the commercially available SphygmoCor System (AtCor Medical LTD, Australia). All measurements were performed while the patient was in a recumbent position at room temperature of 25۫ C, between 06:30 and 08:30 A.M. after an overnight fasting (8-10 hours) and after a short period of rest. Peripheral pressure waveforms were recorded from the radial artery at the wrist, using applanation tonometry with a high fidelity micromanometer. When sequential waveforms were recorded, a validated 16-18 generalized transfer function was applied to generate the corresponding central pressure waveform. The integral system software was used to calculate an average radial artery waveform and to derive a corresponding central aortic pressure waveform using a previously validated generalized transfer function. From these data the indexes of arterial stiffness were obtained. The augmentation of central arterial pressure is the difference between the first and second systolic peaks of the central pressure waveforms, and the central augmentation index (AIx) is the augmentation expressed as a percentage of the pulse pressure.

This technology is easy to perform, non-invasive, simple, rapid (15 minutes per test) and repeatable.

Oxidized LDL Blood samples were collected in EDTA containing tubes. Separation of plasma was performed by centrifugation at 2500 RPM for 10 minutes. In order to neutralize the effect of rheumatoid factor on test accuracy, 5% anti-interference reagent was added to the plasma. Concentration of ox-LDL was determined using an Elisa kit manufactured by Dyne Diagnostic.

Highly sensitive CRP Level was measured using the latex immunonephelometry technique according to manufacturer protocols. Levels were determined with a concentration restriction of 0.0175 mg/dL.

Cholesterol and HDL-cholesterol were measured by standard techniques.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory evidence of subclinical hypothyroidism (TSH levels 4-25 mU/L and normal T4 values) in at least two following tests (one month apart from each other)

Exclusion Criteria:

* Recent (less than 6 months) myocardial infarction, cerebrovascular event or angiography with stent placement
* Serious infection in the month before recruitment
* Any use of contrast media in the last 6 months
* Loss of more than 5% of body weight during the last 6 months
* Cardiac arrhythmias
* Ejection fraction of less than 40%
* Active malignant diseases
* Previous thyroid disease and
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-07; Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Koren, MD, Principal Investigator — Department of Internal Medicine A , Research & Development unit Assaf Harofeh Medical Center, Zerifin, affiliated to Sackler School of Medicine,